CLINICAL TRIAL: NCT06267430
Title: The Effectiveness of a Personalized Executive Functioning Training Program for Pre-schoolers With a Severe Congenital Heart Disease
Brief Title: Learning by Heart: The Effectiveness of an EF Training Program for Pre-schoolers With a Severe CHD
Acronym: LbH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Andre Rietman, Doctor, Neuropsychologist, Erasmus Medical Center
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: NL85141.078.23
Record Dates: First submitted 2023-12-12; First posted 2024-02-20 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Congenital Heart Disease; Executive Dysfunction; Attention Disorder
Keywords: Congenital heart disease; Preschooler; Executive functions; Training
MeSH Terms: conditions — Heart Defects, Congenital; Cognition Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The psychologist testing all participants, will be blinded for the allocation of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants allocated to the intervention group will receive the personalised training program 'KleuterExtra', developed by dr. Lex Wijnroks from Utrecht University. All parents will receive the book 'Speels Brein' ('Playful Brain') and an age-appropriate addition for preschoolers to this book.
  Interventions: Behavioral: Kleuter Extra training program
- Control group (No Intervention): As described, the parents of the control group will also receive the book 'Speels Brein' ('Playful Brain') and the age-appropriate addition for preschoolers to this book.

INTERVENTIONS:
Behavioral: Kleuter Extra training program — The intervention was described in the included arm/group explanation.
  Arms: Intervention group

SUMMARY:
Advances in prenatal and neonatal care have improved outcomes in children with severe congenital heart disease (CHD). With the increase in survival, neurocognitive problems such as executive functioning (EF) impairments have become more apparent in these children. EF problems have cascading negative effects on a child's development. New insights in EF development suggest that in otherwise physically healthy young children, EF can be improved by training. In a pilot study funded by Stichting Hartekind, the investigators studied the feasibility of a personalized EF training program called 'Kleuter Extra' and the results were promising. Therefore, the current study will investigate the effectiveness of this program in 4-6-year-old children with severe CHD. The researchers will also explore interactions between the parent-child relationship and EF development of the child as psychosocial difficulties in these children and their parent(s) and/or caretaker(s) may impact EF-development. If found effective, EF training for children with severe CHD will improve their developmental outcome.

DETAILED DESCRIPTION:
Advances in prenatal and neonatal care have improved outcome in children with severe congenital heart disease (CHD), with survival rates up to 90%. With the increase in survival, neurocognitive problems and psychological maladjustment have become more apparent in these children, such as impairments in their executive functioning. Executive functioning (EF) is an umbrella-term for several higher-order cognitive processes crucial for self-regulated and goal directed behaviour. Frequently postulated components of EF are inhibition, including motor inhibition, and attention, working memory, and cognitive flexibility. Early EF problems often result in emotion regulation difficulties, behavioural problems, social problems, and learning problems, which can lead to diminished functioning in social domains and lower achievement levels in education and employment status. Children with CHD might be rendered even more vulnerable for EF-problems since EF development is embedded within the social context of a child. There is an increasing understanding of how naturally distressing the CHD diagnosis and treatment can be for parents, which can impair the interactions with their child and in turn might negatively impact the child's EF development. Looking at the reciprocal nature of relationships, the child's illness and/or emotional and behavioural problems that may be associated with EF difficulties might negatively impact the parent-child relationship, parenting behaviour and parental wellbeing. However, these relations are poorly understood, especially regarding fathers. A greater understanding of the interplay between biological and psychosocial factors on EF-development is needed to promote optimal developmental outcomes for these vulnerable children.

New insights suggest that EF can be improved by training. Due to neural plasticity, the window for effective training seems to be between the ages of two and six years. After this time frame, improvements in EF may not retain after training or not generalize to off-task functions. Current EF training programs are not personalised ('adaptive') but offer the same program regardless of the specific child's EF dysfunctions, which may explain their limited effects. There is presently no effective EF training program for children with CHD.

In a pilot study funded by Stichting Hartekind, the researchers investigated the feasibility of a personalised EF training program called 'KleuterExtra' in 4-6 year old children with severe CHD. Within a week, 31 children were (self-) referred for the study, indicating a great clinical need. Directly after training, children showed clinically relevant improvement on the specific EFs targeted in training, with Cohen's d effect sizes ranging from 0.19 to 2.41 (>1.00 on 5 out of 9 tasks). Improvement was also found in untrained EFs and tasks that combined multiple EFs, indicating a generalization effect. Parents and teachers spontaneously reported positive results in daily life. Based on these promising results, the investigators designed the current randomized, controlled study to test the effectiveness of this training program in pre-schoolers with severe CHD.

Given the above, the investigators designed this study to investigate the effectiveness of a tailored EF training program for preschoolers with severe CHD. Secondary aim was to explore interactions between the parent-child relationship and the EF development of the child. If found effective, EF training for children with severe CHD will improve their developmental outcome.

ELIGIBILITY:
In order to be eligible to participate in this study, a child must meet all of the following criteria:

* Aged 4.0 - 6.0 years upon inclusion OR aged 6.0-7.0 years who are still in kindergarten (group 1 & 2 of the Dutch school system)
* Required CHD surgery in the first six months of life (with or without ECMO) or a cyanotic CHD that required surgery in the first 12 months of life
* IQ estimated > 55 (no moderate to severe intellectual disability)
* Diminished EF based on a below average score on any of the subtests of the 'KleuterExtra' test battery (≤ 25 percentile) at t = 0
* Sufficient comprehension of the Dutch language by the child to be able to participate in the EF test battery and the EF training program. In order to be eligible to participate in this study, the parent(s) must meet the following criteria:
* Sufficient comprehension of the Dutch language to understand the study information and to be able to fill out the Dutch questionnaires.

Exclusion Criteria:

* Children receiving targeted EF support at school upon inclusion.
* Children with severe brain damage (estimated IQ < 55)
* Genetic syndromes known to directly affect cognitive performance (e.g. Down syndrome)
* Children with severe psychiatric disorders upon inclusion that require treatment first, such as a posttraumatic stress disorder, separation anxiety disorder, or reactive attachment disorder.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-11-02 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Kleuter Extra test battery | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  The primary endpoint is a single composite score on the 'Kleuter Extra' EF test battery. This composite score will be statistically derived from the individual test results of the test battery. Therefore, the minimum and maximum values cannot be provided at this point, nor whether a higher score means a better or worse outcome.

SECONDARY OUTCOMES:
EF functioning | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  Single test scores from the ''Kleuter Extra'' EF test battery:
  * subtest 'Pencil Tap'. Scores range from 0 to 100.
  * subtest 'Go/No go animals'. Scores range from 0 to 60.
  * subtest 'Statue task'. Scores range from 0 to 30.
  * subtest 'Search task'. Scores range from 0 to 35.
  * subtest 'Sustained attention'. Scores range from 0 to 30.
  * subtest 'Corsi blocks'. Scores range from 0 to 26.
  * subtest 'Dots'. Scores range from 0 to 37.
  * subtest 'Numbers'. Scores range from 0 to 54.
  * subtest 'Three is Correct'. Scores range from 0 to 78.
  * subtest 'Head-Shoulders-Knees-Toes'. Scores range from 0 to 52.
  A higher score indicates a better outcome for all subtests, except the 'Pencil Tap' task.
  The scores are converted into percentiles ranging from the lowest percentile rank (0-3) to the highest percentile rank (>75) with a higher score indicating a better outcome.
Information processing | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  Cognitive Proficiency Index of the WPPSI-IV-NL. This index score is based on the test results of the following subtests:
  * subtest 'Picture Memory'
  * subtest 'Zoo Locations'
  * subtest 'Bug Search'
  * subtest 'Cancellation'
  * subtest 'Animal Coding'. The scale scores range from 1 to 19 and a higher score indicates a better outcome.
Executive functioning in daily life - completed by the parent(s) | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  Behavior Rating Inventory of Executive Function - Preschool Version questionnaire (BRIEF-P): t-scores range from 20-80, higher scores indicate worse outcome)
Behavioral and emotional difficulties of the child - completed by the parent(s) | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  Child Behavioral Checklist questionnaire 1,5 - 5 years old (CBCL): t-scores range from 50-100, higher scores indicate worse outcome)
Quality of the child's life - completed by the parent(s) | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  Preschool Children Quality of Life questionnaire (TAPQOL): t-scores range from 0 - 100, higher score indicates better outcome.
Emotional distress parent - completed by the parent(s) | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  Depression, Anxiety, Stress Scale (DASS-21): scores range from 0-63, higher score indicates worse outcome)
Parental trauma | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  PCL-5 questionnaire ('PCL-5' is the title, scores range from 0-80, higher score indicates worse outcome)
Parenting behavior and quality parent-child relationship - completed by the parent(s) | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  Parenting Behavior questionnaire (PABI): scores range from 0-525, a higher score can mean a better or worse outcome depending on the specific scale.
Child demographics teacher's perspective | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  Additional support in school, type, being held back a year (qualitative data, designed by the study group)
Behavioral and emotional difficulties teacher's perspective | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  Teacher's Report Form questionnaire (TRF): t-scores range from 50-100, higher scores indicate worse outcome)
Executive functioning child in daily life teacher's perspective | 9 weeks after baseline. Additional measures at 6 months and 12 months after baseline.
  Behavior Rating Inventory of Executive Function questionnaire - teachers (BRIEF); t-scores range from 20-80, higher scores indicate worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: André Rietman, Principal Investigator — Erasmus Medical Center; Renske Schappin, Principal Investigator — Erasmus Medical Center
Locations (3):
- Netherlands (3):
  - University Medical Center - Beatrix children's hospital Groningen, Groningen
  - Erasmus Medical Center Sophia Children's Hospital, Rotterdam
  - University Medical Center - Wilhelmina children's hospital Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No